CLINICAL TRIAL: NCT00355693
Title: Effect Site Controlled, Reaction Time Safeguarded, Patient Maintained Sedation With Propofol A) in Oral Surgery Patients B) in General Dentistry Patients C) in Colonoscopy Patients
Brief Title: Effect Site Controlled, Reaction Time Safeguarded, Patient Maintained Sedation With Propofol in Anxious Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Equity Partners (University Challenge Fund) (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9812/A
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2006-08-24 (Estimated); Status verified 2006-04

CONDITIONS: Oral Surgical Procedures; Surgery, Oral; Dental Anxiety; Surgery; Colonoscopy
Keywords: Anxiety; Dental; Oral; Surgery; Colonoscopy; Propofol; Sedation; Effect; Reaction
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Device: Pump for propofol delivery

SUMMARY:
Whether patient-maintained sedation (the patient controls his/her degree of sedation using a hand-held device) using the drug propofol is safer and more effective when using deteriorating reaction time as an added safeguard against the potential for over sedation in a groups of patients undergoing oral surgery, general dentistry and colonoscopy.

DETAILED DESCRIPTION:
Patients receiving conscious sedation for dentistry and endoscopy are usually treated with intermittent bolus doses of intravenous midazolam (administered by the operator-sedationist). The safety of such a regime has been questioned with reports of up to 13 % of patients desaturating to below 80 % in the recovery area following sedation for endoscopy. Mortality occurs in 0.05 % of endoscopy patients (with approximately 60 % of this being due to hypoxaemia). The aim of our work, therefore, is to look at providing sedation that is both safer as well as being efficacious.

The drug propofol, the agent most commonly used to induce general anaesthesia in the UK, is also frequently administered intravenously by anaesthetists in low doses to provide conscious sedation for patients undergoing unpleasant procedures i.e. patients become relaxed, anxiety-free, but maintain verbal contact throughout.

The technique of patient maintained sedation using the drug propofol (the patient can increase the amount of sedation (and propofol) they receive by pressing a demand button attached to a standard infusion device) has been used by anaesthetists and evaluated since 1997.

Several recent studies published and submitted for publication by this research group on patient maintained sedation using the drug propofol have shown this method of sedation to be safe and effective in dental patients (over 120 patients studied). It was also shown that this method, when compared to the established method of sedation in oral surgery (the dentist administering doses of midazolam intravenously), to produce both quicker recovery and less anxiety prior to the surgery.

The routine use of propofol traditionally is restricted to anaesthetists, as in high doses general anaesthesia is produced with possible loss of airway patency. Currently the safety feature is predominantly that as patients become more sedated they cannot press the patient demand button and hence cannot increase the amount of propofol they are receiving. Also the device ensures that the blood and brain concentrations have equilibrated to within 10% of each other before another successful demand for propofol can be made (usually takes approximately two minutes) and it only allows a maximum calculated brain concentration of 3 micrograms/milliliter of propofol. The device also will start to decrease the calculated brain concentration of propofol if the demand button has not been pressed for six minutes.

Despite the encouraging results above we also found in a recent pilot study involving 20 healthy volunteers who were instructed to try and make themselves unconscious that there were 2 cases of over sedation (of these one briefly lost verbal contact and the other required supplemental oxygen only). Over sedation, however, was not demonstrated with any of the oral surgery patients in the previous studies. This may have been due to a higher level of anxiety in dental patients affecting response to propofol.

We have therefore incorporated an additional safety feature into the existing and previously studied patient maintained sedation system which may further decrease or eliminate this small risk of over sedation. All the above safety features are retained and in addition the patient demand button will now also be used to monitor reaction time at one minutely intervals.

It is known that propofol slows the reaction time of a given individual and in another recent study of 40 patients undergoing general anaesthesia for planned surgery using propofol, the patients' reaction times were recorded both awake and during induction of anaesthesia by instructing the patients to press a button as quickly as possible in response to the handset vibrating. The calculated effect site (brain) concentration of propofol was increased incrementally and reaction time monitored at each stage until the patient could no longer press the button.

The data from this study (deteriorating patient reaction time with increased brain concentration of propofol) was analysed and this information used to provide an additional safety feature within the system to prevent over sedation i.e. a patient's reaction time deterioration by a certain percentage will prevent himself or herself being able to self-administer more propofol. Furthermore the system will actually start to decrease the brain concentration of propofol once the patients' reaction time becomes too slow. The patient demand button will be used to monitor reaction time at one minutely intervals as well as administer more propofol.

.

We hope that this will eliminate the small risk of over sedation and wish to conduct pilot studies to assess the safety and efficacy of this reaction time safeguarded, patient-maintained sedation system in three groups of twenty patients requiring sedation for planned procedures.

We have chosen two groups of dental patients, one group having oral surgery (technically more difficult dental work e.g. wisdom tooth removal) and one group having routine dentistry (e.g. patients having tooth fillings who are referred for sedation due to high anxiety levels). Another of our outcome measures will look at the effect of this technique on the patients' anxiety levels and we believe that this technique may be beneficial in reducing anxiety levels.

Patient maintained sedation has also been studied in 20 colonoscopy patients and found to be efficacious. However there were also 4 cases of slight over sedation, none of whom required any intervention e.g. airway or circulatory. We hope that by incorporating the reaction time safeguard that we can again eliminate this small risk.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II (healthy or mild systemic illness) undergoing planned dental surgery or colonoscopy.
* Age 18 - 65

Exclusion Criteria:

* ASA III or above
* Out with age group above
* Contraindication to propofol
* History of epilepsy
* History of substance abuse
* Major Psychiatric illness
* Pregnancy or breastfeeding
* Unable or unwilling to give informed consent
* Unable to use necessary apparatus
* Vulnerable groups

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-10; Study Completion 2007-02

PRIMARY OUTCOMES:
Minimal Sedation Level obtained (modified Objective Observers's Assessment of Sedation)
(Scores 5, fully awake to 1, unresponsive)
Maximal change in oxygen saturation (SpO2)

SECONDARY OUTCOMES:
Effect site concentrations of propofol
Anxiety Levels
Requirement for supplementary oxygen (if SpO2 < 90%)
Requirement for airway support
Maximal change in heart rate (HR) and blood pressure (BP)
Operator assessment (ease of procedure, cooperation)
Patient Satisfaction and recollection

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Allam, MB ChB FRCA, Principal Investigator — University of Glasgow Dept of Anaesthesia; Conor P O'Brien, BDS FDS, Principal Investigator — Glasgow Dental Hospital & School; Avril Macpherson, MFDS MSND, Principal Investigator — NHS Lothian
Locations (2):
- United Kingdom (2):
  - Glasgow Dental Hospital and School, Glasgow, Glasgow
  - Duncan Street Dental Centre, Edinburgh